CLINICAL TRIAL: NCT00769327
Title: Front-line Treatment of Philadelphia Positive (Ph Pos), BCRABL Positive, Chronic Myeloid Leukemia (CML) With Two Tyrosine Kinase Inhibitors (TKI) (Nilotinib and Imotinib) A Phase II Exploratory Multicentric Centre.
Brief Title: Nilotinib and Imatinib Mesylate in Treating Patients With Early Chronic Phase Chronic Myelogenous Leukemia
Acronym: CML0408
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CML0408; GIMEMA-CML0408; EUDRACT-2008-004384-19; EU-20881
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Leukemia
Keywords: chronic myelogenous leukemia, BCR-ABL1 positive; chronic phase chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — Imatinib Mesylate; nilotinib; Cytogenetic Analysis; In Situ Hybridization, Fluorescence; Microarray Analysis; Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: imatinib mesylate
Drug: nilotinib
Genetic: cytogenetic analysis
Genetic: fluorescence in situ hybridization
Genetic: microarray analysis
Genetic: mutation analysis
Genetic: polymerase chain reaction
Genetic: polymorphism analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Nilotinib and imatinib mesylate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well giving nilotinib together with imatinib mesylate works in treating patients with early chronic phase chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the complete cytogenetic response rate at 12 months in patients with Philadelphia chromosome- and BCR-ABL-positive early chronic phase chronic myelogenous leukemia treated with nilotinib and imatinib mesylate.

Secondary

* To assess the complete cytogenetic response rate at 6 and 24 months in these patients.
* To assess the major and complete molecular response rate at 6, 12, and 24 months in these patients.
* To assess the frequency and the types of BCR-ABL kinase domain mutations at 24 months during and for 3 years after study treatment.
* To assess the rate of failures and the time to failure at 12, 24, and 60 months in these patients.
* To assess compliance, toxicity, and adverse events in these patients.
* To understand the relationship between response, gene expression profile, biomarkers, and drug plasma concentrations in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral nilotinib twice daily in months 1-3, 7-9, 13-15, and 19-21 and oral imatinib mesylate once daily in months 4-6, 10-12, 16-18, and 22-24. Treatment continues for 24 months in the absence of disease progression or unacceptable toxicity. Patients may be eligible to continue oral nilotinib and oral imatinib mesylate for up to another 36 months if it is in the interest of the patient.

Blood samples and bone marrow biopsies are collected periodically for cytogenetic response by chromosome banding analysis and FISH analysis; real-time quantitative PCR mutational analysis and single nucleotide polymorphism analysis of BCR-ABL transcripts; and gene expression profiling and correlative biomarker studies.

After completion of study therapy, patients are followed every 6 months for 3 years and then every 12 months for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytologically and cytogenetically confirmed chronic myelogenous leukemia meeting the following criteria:

  * Early chronic phase disease (< 6 months from diagnosis)
  * Philadelphia chromosome-positive disease
  * BCR-ABL-positive

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* ALT and AST = 2.5 times upper limit of normal (ULN) (5.0 times ULN if considered due to leukemia)
* Alkaline phosphatase = 2.5 times ULN (unless considered due to leukemia)
* Serum bilirubin = 1.5 times ULN
* Serum creatinine = 1.5 times ULN
* Serum amylase = 1.5 times ULN
* Serum lipase = 1.5 times ULN
* Normal serum levels of the following or correctable with supplements:

  * Potassium
  * Total calcium (corrected for serum albumin)
  * Magnesium
  * Phosphorus
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier method contraception during study and for up to 3 months following completion of study treatment
* No impaired cardiac function, including any of the following:

  * LVEF < 45% by MUGA scan or echocardiogram
  * Uncontrolled congestive heart failure
  * Uncontrolled hypertension
  * Uncontrolled angina pectoris
  * Myocardial infarction within the past 12 months
* No significant electric heart abnormalities, including any of the following:

  * History or active ventricular or atrial tachyarrhythmias
  * Congenital long QT syndrome and/or QTc > 450 msec on screening ECG
* No history of acute (within one year) or chronic pancreatitis
* No impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* No acute or chronic liver or renal disease considered unrelated to leukemia
* No known diagnosis of HIV infection
* No other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes, active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol
* No other primary malignancy that is currently clinically significant or requires active intervention

PRIOR CONCURRENT THERAPY:

* More than 2 weeks since prior major surgery and recovered
* More than 30 days since prior imatinib mesylate, with a washout period of ≥ 7 days
* More than 4 weeks since prior investigational drug
* No prior hematopoietic stem cell transplantation
* No concurrent therapeutic coumarin derivates (i.e., warfarin, acenocoumarol, phenprocoumon)
* No concurrent medications that would prolong the QT interval
* No concurrent chemotherapy, investigational agents, radiotherapy, or biologic therapy
* Prior treatment with hydroxyurea or anagrelide allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2009-02-09 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10-10 (Actual)

PRIMARY OUTCOMES:
Complete cytogenetic response rate | At 12 months from study entry

SECONDARY OUTCOMES:
Complete cytogenetic response | At at 6 and 24 months from study entry
Major and complete molecular response rate | At at 6, 12 and 24 months from study entry
Development of BCR-ABL kinase domain mutations (number, timing, and type) | At at 24 months during and for 3 years after study treatment
Rate of failures and the time to failure | At 12, 24, and 60 months from study entry
Safety and tolerability | At 24 months from study entry
Frequency and type of adverse events (AE) and severe AE | At 24 months from study entry
Relationship between response, the gene expression profile, the biomarkers of leukemic cells, and plasma concentrations of nilotinib and imatinib mesylate | At 24 months from study entry

CONTACTS AND LOCATIONS:
Overall Officials: Michele Baccarani, MD, Principal Investigator — Gruppo Italiano Malattie EMatologiche dell'Adulto
Locations (37):
- Italy (37):
  - Centro Oncologico Basilicata, Rionero in Vulture, Potenza
  - Ospedale Civile Alessandria, Alessandria
  - Dipartimento Area Medica P.O., Ascoli Piceno
  - S.G. Moscati Hospital, Avellino
  - Unità Operativa Ematologia 1 - Università degli Studi di Bari, Bari
  - Ospedali Riuniti di Bergamo, Bergamo
  - Ist.Ematologia e Oncologia Medica L.e A. Seragnoli, Bologna
  - ASL N.8 - Ospedale "A. Businco" - Struttura Complessa di Ematologia e CTMO, Cagliari
  - Ctc U.O Di Ematologia Con Trapianto Di Midollo Osseo - Catania, Catania
  - Unità di Oncoematologia Azienda Ospedaliera Garibaldi, Catania
  - Azienda Ospedaliera Pugliese Ciaccio - Presidio Ospedaliero A.Pugliese - Unità Operativa di Ematologia, Catanzaro
  - Sez.Ematologia e Dip. scienze Biomediche Arcispedale S. Anna, Ferrara
  - Azienda Ospedaliera di Firenze, Florence
  - Struttura Complessa di Ematologia Ospedali Riuniti Foggia - Azienda Ospedaliero-Universitaria, Foggia
  - Clinica Ematologica - DiMI - Università degli Studi di Genova, Genova
  - Clinica Ematologica - Università degli Studi, Genova
  - A.O. Universitaria Policlinico Martina di Messina, Messina
  - Azienda ospedaliera Ospedali Riuniti "Papardo Piemonte", Messina
  - Sez. di medicina Interna Oncologia ed Ematologia, Modena
  - Universtià degli Studi di Napoli "Federico II" - Facoltà di medicina e chirurgia, Napoli
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Dip. di Scienze Cliniche e Biologiche - Ospedale S. Luigi Gonzaga, Orbassano
  - Ospedali Riuniti "Villa Sofia-Cervello", Palermo
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Unità Operativa Ematologia e Centro Trapianti - Dipartimento di Oncologia ed Ematologia - AUSL Ospedale di Piacenza, Piacenza
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Unità operativa complessa di Ematologia, Reggio Emilia
  - A.O Umberto I, Roma
  - Complesso Ospedaliero S. Giovanni Addolorata, Roma
  - Ospedale S.Eugenio, Roma
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - U.O. Ematologia, Azienda Ospedaliera Universitaria Senese, Siena
  - Azienda ospedaliera S. Maria di Terni, Terni
  - SCDO Ematologia 2 AOU S.Giovanni Battista, Torino
  - Policlinico Universitario Udine, Udine
  - Policlinico G. B. Rossi - Borgo Roma, Verona
  - Ospedale San Bortolo, Vicenza

REFERENCES:
- [Derived] Castagnetti F, Gugliotta G, Baccarani M, Breccia M, Specchia G, Levato L, Abruzzese E, Rossi G, Iurlo A, Martino B, Pregno P, Stagno F, Cuneo A, Bonifacio M, Gobbi M, Russo D, Gozzini A, Tiribelli M, de Vivo A, Alimena G, Cavo M, Martinelli G, Pane F, Saglio G, Rosti G; GIMEMA CML Working Party. Differences among young adults, adults and elderly chronic myeloid leukemia patients. Ann Oncol. 2015 Jan;26(1):185-192. doi: 10.1093/annonc/mdu490. Epub 2014 Oct 30. PMID 25361995